CLINICAL TRIAL: NCT04430335
Title: Cultural and Linguistic Adaptation of a Telephone-Based Intervention to Treat Depression and Anxiety in Hispanic Cancer Survivors
Brief Title: Telephone-Based Intervention to Treat Depression and Anxiety in Hispanic Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00066444; WFBCCC 01220 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Survivorship; Cancer; Depression, Anxiety
MeSH Terms: conditions — Neoplasms; Depression; Anxiety Disorders | interventions — Interviews as Topic; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telephone-Based Cognitive Behavioral Therapy (Other): Participants with moderate or severe anxiety and/or depressive symptoms will participate in the telephone-based intervention that consists of the CBT workbook (15 minutes daily to complete exercises), plus psychotherapy delivered by telephone with a licensed bilingual mental health provider (45-50 minute sessions weekly).
  Interventions: Behavioral: Telephone interview; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Telephone interview — Interested participants will complete a telephone interview to determine eligibility for the study. If found to be eligible for the study, participants will be registered and set up a time to speak with an assigned study coach.
Behavioral: Cognitive Behavioral Therapy — Participants will speak with their assigned coach over the phone for 12 weeks to discuss the cognitive behavioral therapy (CBT) study workbook and provide feedback. CBT is a type of treatment that teaches people different ways to handle anxiety and/or depressive symptoms, such as by relaxing the body, changing thoughts, and solving problems. Participants will receive a workbook focused on teaching these strategies.

SUMMARY:
The purpose of this research is to assess the feasibility of administering a telephone-based intervention to treat depression and anxiety in Hispanic cancer survivors.

DETAILED DESCRIPTION:
Primary Objectives

* To assess the feasibility (participation, accrual, retention, adherence) of administering the intervention in Hispanic cancer survivors.
* To culturally adapt an existing behavioral intervention for cancer survivors based on stakeholder feedback.

Exploratory Objectives

* To summarize emotional distress (anxiety, depressive symptoms) and fear of recurrence in these post-treatment Hispanic cancer survivors.
* To describe the therapy process in terms of satisfaction with treatment and the therapist-participant relationship.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion: age greater than or equal to 18 years;
* Self-identify as Hispanic ethnicity
* Score greater than or equal to 10 on the General Anxiety Disorder (GAD)-7 and/or greater than or equal to 8 on the Patient Health Questionnaire (PHQ)-9
* History of (1) treated (newly diagnosed or recurrent) solid tumor cancers (Stage I, II, or III); (2) any stage lymphoma (Hodgkin's or non-Hodgkin's); (3) acute leukemia in remission for more than a year; (4) chronic myelogenous leukemia with stable disease (chronic phase disease); or (5) chronic lymphocytic leukemia (CLL) not requiring treatment or a change in treatment for more than 6 months.
* 6-60 months post-treatment (surgery, chemotherapy, and/or radiation therapy) for cancer (If only received active surveillance for prostate cancer or lymphoma with no other cancer treatment, participant is ineligible.) The timeframe applies to the most recent completion of treatment if a participant had a cancer recurrence. It is acceptable to be on hormonal/maintenance therapies.
* Must be able to speak, read, and understand Spanish or English.
* Resides in North Carolina.

Exclusion Criteria:

* Current psychotherapy [regular appointment(s) with a mental health provider within the last 30 days]
* Self-reported active alcohol or substance abuse within the last 30 days
* Past history of prostate cancer or non-Hodgkin's lymphoma with only active surveillance (i.e., no surgery, chemotherapy, or radiation therapy)
* Progressive cancer
* Global cognitive impairment based on self-reported diagnosis of dementia.
* Self-reported psychotic symptoms in the last 30 days (Item in Screening Form: "Have you seen things that aren't really there or have you heard voices when no one else was around within the last 30 days?")
* Active suicidal ideation with plan and intent
* Any change in psychotropic medications within the last 30 days
* Hearing loss that would preclude participating in telephone sessions (determined by brief hearing assessment administered by research staff). Individuals who can compensate for hearing loss through the use of a hearing device or TDD phone, and through the use of such devices are able to communicate with the study therapist by telephone, will be included. If the therapist cannot communicate with the participant by telephone, the participant will be excluded.
* Failure/inability/unwillingness to provide names and contact information for two family members or friends to serve as emergency contacts during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C Danhauer, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Origin of Ethnicity - Mexico | 5
  Origin of Ethnicity - Honduras | 1
  Origin of Ethnicity - Nicaragua | 1
  Origin of Ethnicity - Spain | 1
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Participation Rate - Percentage Who Agreed to Participate
Description: To determine participation rate, investigators will track the total number of individuals approached, the number of individuals who met all eligibility criteria and percent who agree to participate.
Time Frame: 12 weeks after start of intervention
Measure: Number; unit: percentage of participants
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
percentage of participants | 88.9

2. Primary Outcome: Accrual Rate
Description: Accrual rates will be calculated by calculating the mean number of participants recruited per month.
Time Frame: 12 weeks after start of intervention
Measure: Number; unit: participants accrued per month
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
participants accrued per month | 1.1

3. Primary Outcome: Retention Rate - Percentage of Completed Visits
Description: Study retention will be estimated by the proportion of participants who complete the Week 13 visit. Drop-out is defined as 100% minus the dropout %
Time Frame: 13 weeks after the start of intervention
Measure: Number; unit: percentage of completion of Wk. 13 visit
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
percentage of completion of Wk. 13 visit | 87.5

4. Primary Outcome: Adherence - Percentage of Completed Therapy Sessions
Description: Intervention adherence will be estimated as the mean percentage of therapy or check-in sessions each participant completes. Participants must complete at least 9 of the 12 sessions (75%) to be considered adherent.
Time Frame: 12 weeks after start of intervention
Measure: Number; unit: percentage to complete 9 or more session
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
percentage to complete 9 or more session | 87.5

5. Secondary Outcome: Anxiety Questionnaire - General Anxiety Disorder (GAD)-7
Description: The General Anxiety Disorder (GAD)-7 is a self-report measure of DSM-IV symptoms of general anxiety disorder. Participants rate 7 questions on a scale of 0 (not at all), 1 (several days), 2 (more than half the days) and 3 (nearly every day); one additional question assesses the interference of these symptoms with functioning. The first 7 questions are summed to create a total score. Scoring range is 0-21 with the higher score indicating a higher level of anxiety (scores 0 to less than or equal to 9 = no/mild anxiety; scores greater than or equal to 10 to less than or equal to 14 = moderate anxiety; scores greater than or equal to 15 to 21 = severe anxiety).
Time Frame: At baseline, 7 weeks and 13 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
score on a scale
  Baseline | 12.9 (2.0)
  Week 7 | 4.3 (2.3)
  Week 13 | 4.1 (2.1)

6. Secondary Outcome: Depressive Symptoms Questionnaire - Patient Health Questionnaire (PHQ)-9
Description: The Patient Health Questionnaire (PHQ)-9 is a self-report measure of DSM-IV symptoms of Major Depressive Disorder. Participants rate how often they have experienced nine symptoms over the past 2 weeks on a scale of 0 (not at all); 1 (several days), 2 (more than half the days) and 3 (nearly every day). Responses are summed, with higher scores indicating greater depressive symptomatology. Scoring scale = 0-27 (scores 0 to less than or equal to 7 = no/mild depressive symptoms; scores greater than or equal to 8 to less than or equal to 14 = moderate depressive symptoms; scores greater than or equal to 15 to 27 = severe depressive symptoms)
Time Frame: At baseline, 7 weeks and 13 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
score on a scale
  Baseline | 11.9 (2.0)
  Week 7 | 4.3 (2.3)
  Week 13 | 4.1 (2.1)

7. Secondary Outcome: Fear of Cancer Recurrence Inventory Questionnaire
Description: The Fear of Cancer Recurrence Inventory (FCRI; severity subscale) will be used to measure self-reported fear of recurrence. This 9-item subscale measures the presence and severity of the intrusive thoughts or images associated with the fear of recurrence. Scoring scale ranges from 0 (not at all or never) to 4 (a great deal or all of the time). Score ranges from 0-36. The higher the score, the greater the participants' fear of recurrence.
Time Frame: At baseline and 13 weeks after start of intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 7
score on a scale
  Baseline | 15.5 (3.1)
  Week 13 | 11.6 (3.3)

ADVERSE EVENTS:
Time Frame: 7 weeks after the start of study intervention and again at 12 weeks after the start of study intervention.
Arm/Group | Telephone-Based Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT04430335/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT04430335/ICF_000.pdf